CLINICAL TRIAL: NCT02871609
Title: Longterm Ureteral Stenting: Assessment of Stent- Associated Morbidity, Associated Costs and Impact of Biofilms
Brief Title: Assessment of Longterm Ureteral Stenting
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Patrick Betschart, Dr. med., Cantonal Hospital of St. Gallen
Other Study IDs: CTU 16.011
Record Dates: First submitted 2016-08-05; First posted 2016-08-18 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Longterm Indwelling Ureteral Stent
Keywords: Biofilm; Morbidity; Ureteral Catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with longterm ureteral stent
  Interventions: Other: Stent examination, urinary analysis, USSQ questionnaire

INTERVENTIONS:
Other: Stent examination, urinary analysis, USSQ questionnaire

SUMMARY:
This study is performed to analyze various aspects of biofilms on ureteral stents in a longterm setting.

DETAILED DESCRIPTION:
The study is performed to provide a better understanding of the influence of biofilms on ureteral stents on the entire spectrum of stent-associated morbidity in a longterm setting.

In addition, the trial is intended to give an overview of the incidence of complaints, the occurrence of complications and their economic aspects.

The influence of biofilms on the morbidity associated with longterm ureteral stenting is assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with longterm indwelling ureteral stent (minimum of 2 months) undergoing regular changes
* Informed consent
* responsible patients

Exclusion Criteria:

* ongoing therapy: OAB, LUTS, urinary incontinence, chronic prostatitis, chronic pelvic pain syndrome
* insufficient language skills
* cognitive limitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with longterm indwelling ureteral stent undergoing regular changes in an inpatient or outpatient setting at the department of urology of KSSG.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2016-07; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Total biofilm mass on ureteral stents | Time of stent removal/change: three months (range 2-4 months) after last stent insertion/change
Assessment of morbidity using the Ureteral Stent Symptom Questionnaire (USSQ) | Day of stent removal/change: three months (range 2-4 months) after last stent insertion/change

SECONDARY OUTCOMES:
Urine Culture | 2-6 months after stent insertion
Number of bacteria on stent surface, if applicable number of bacteria on two indwelling stents | 2-6 months after stent insertion
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2-6 months after stent insertion
Assessment of costs arising from complications | 2-6 months after stent insertion
  complications assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Betschart, Dr. med., Principal Investigator — Department of Urology
Locations (1):
- Urological Department, Cantonal Hospital of St. Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No